CLINICAL TRIAL: NCT05881122
Title: The Effects of an Anti-inflammatory Dietary Consultation on Self-efficacy, Adherence and Selected Health Outcomes: A Randomized Control Trial
Brief Title: Anti-inflammatory Diet Consultation for Those With Neuromuscular Disability
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brock University (Other)
Responsible Party: Principal Investigator, David Ditor, Professor, Brock University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 21-054 - Ditor
Record Dates: First submitted 2023-04-17; First posted 2023-05-31 (Actual); Last update posted 2023-05-31 (Actual); Status verified 2023-05

CONDITIONS: Inflammation; Spinal Cord Injuries; Multiple Sclerosis; Muscular Dystrophies; Diet Habit
MeSH Terms: conditions — Inflammation; Spinal Cord Injuries; Multiple Sclerosis; Muscular Dystrophies; Feeding Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mad Dog Dietary Consultation Intervention group (Experimental): The intervention group received recipes for an anti-inflammatory diet and the 2-part consultation. The consultation consisted of a home-visit that included cooking and accessible kitchen equipment demonstrations, and an accompanied trip to the grocery store.
  Interventions: Behavioral: Mad Dog Dietary Consultation
- Control group (No Intervention): The controls received the recipes only.

INTERVENTIONS:
Behavioral: Mad Dog Dietary Consultation — The Mad Dog consultation was delivered in two parts over consecutive days. Part I entailed an accompanied trip to the participant's preferred grocery store to show the participant where selected foods could be found, how to read nutrition labels so that acceptable substitutions to the Mad Dog ingredients could be made, and how to shop for value when choices are presented. Part II of the consultation occurred in the participant's home and focused on meal preparation and kitchen accessibility, as well as a brief overview regarding the negative consequences of chronic inflammation, and the positive effects of adopting an anti-inflammatory diet. Questions and discussion were highly encouraged throughout the consultation and materials were left with the participants allowing them to easily review and reference information that was covered during the meeting. Specifically, participants were given 28 compliant recipes, additional snack ideas and shopping tips along with a consult summary.
  Arms: Mad Dog Dietary Consultation Intervention group

SUMMARY:
This study investigated the effects of a 2-part dietary consultation on adherence to an anti-inflammatory diet in individuals with neuromuscular disability. The effects on self-efficacy for adhering to the diet as well as neuropathic pain and depression one month post-consult were also determined.

DETAILED DESCRIPTION:
This study investigated the effects of a 2-part dietary consultation (the Mad Dog consult) on adherence to an anti-inflammatory diet (the Mad Dog diet) in individuals (N=11) with spinal cord injury, multiple sclerosis and muscular dystrophy. participants were randomly allocated into either the intervention group (n=7) or the control group (n=4).

The Mad Dog consultation was delivered in two parts over consecutive days. Part I entailed an accompanied trip to the participant's preferred grocery store in order to show the participant where selected foods could be found, how to read nutrition labels so that acceptable substitutions to the Mad Dog ingredients could be made, and how to shop for value when choices are presented. Part II of the consultation occurred in the participant's home and focused on meal preparation and kitchen accessibility, as well as a brief overview regarding the negative consequences of chronic inflammation, and the positive effects of adopting an anti-inflammatory diet. Accordingly, the researchers traveled to the participant's home and prepared two sample dinner meals for the participant in an interactive and instructional format. The researchers also brought selected pieces of accessible cooking equipment (designed for use in those with reduced hand function) which were demonstrated during the meal preparation. Participants were not given the equipment to keep, but they were instructed where to buy the equipment online if they found it beneficial. Questions and discussion were highly encouraged throughout the consultation and materials were left with the participants allowing them to easily review and reference information that was covered during the meeting. Specifically, participants were given a booklet with 28 compliant recipes, additional snack ideas and shopping tips along with a brochure summarizing the consult. The combined length of the consult was approximately 90-120 minutes.

Lastly, the Mad Dog consultation also included a virtual group, where participants could share and discuss anti-inflammatory recipes (that may complement the recipes in the Mad Dog diet) and engage in social support. Researchers were part of the group to oversee discussion but did not participate.

The control group only received the Mad Dog diet recipes, but did not take part in the consultation.

Adherence to the Mad Dog diet was determined by 7-day food logs before the intervention and at one month post-intervention. Task and barrier self-efficacy were determined by questionnaire at baseline (immediately after viewing the Mad Dog Diet), immediately after the consultation (in the intervention group only ) and at one month post-intervention (in both groups). Neuropathic pain and depression were determined by the Neuropathic Pain Questionnaire and the Centre for Epidemiological Studies Depression (CES-D) questionnaire at baseline and at one month post-intervention (in both groups).

ELIGIBILITY:
Inclusion Criteria:

* To be eligible for this study, participants were required to be over 18 years of age, fluent in English and at least one year removed from either SCI or neurological diagnosis. All participants but one (who had muscular dystrophy) had either spinal cord injury (SCI) or multiple sclerosis (MS). Participants with SCI could have any level or severity of injury while participants with MS could have had any type of MS.

Exclusion Criteria:

* Younger than 18
* Not fluent in English
* No SCI or diagnosis of MS or muscular dystrophy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-05-30 (Actual)

PRIMARY OUTCOMES:
Custom-designed task self-efficacy questionnaire | Baseline (for the intervention group and the control group)
  Confidence in one's abilities to adhere to the anti-inflammatory diet. This is a 6-item questionnaire that asks how confident participants are about adhering to the diet for certain amounts of time at certain amounts at certain percentages of adherence. Each item is scored from 1 (not confident at all) to 7 (completely confident). The minimum score is 6 and the maximum score is 42, and higher scores indicate greater self-efficacy.
Custom-designed task self-efficacy questionnaire | Immediately post-intervention (in the intervention group only)
  Confidence in one's abilities to adhere to the anti-inflammatory diet. This is a 6-item questionnaire that asks how confident participants are about adhering to the diet for certain amounts of time at certain amounts at certain percentages of adherence. Each item is scored from 1 (not confident at all) to 7 (completely confident). The minimum score is 6 and the maximum score is 42, and higher scores indicate greater self-efficacy.
Custom-designed task self-efficacy questionnaire | One month post-intervention (for the intervention group and the control group)
  Confidence in one's abilities to adhere to the anti-inflammatory diet. This is a 6-item questionnaire that asks how confident participants are about adhering to the diet for certain amounts of time at certain amounts at certain percentages of adherence. Each item is scored from 1 (not confident at all) to 7 (completely confident). The minimum score is 6 and the maximum score is 42, and higher scores indicate greater self-efficacy.
Custom-designed barrier self-efficacy questionnaire | Baseline (for the intervention group and the control group).
  Confidence in one's ability to overcome the barriers associated with adhering to anti-inflammatory diet. This is a 7-item questionnaire that asks participants how confident they are about overcoming the barriers associated with adhering to the anti-inflammatory diet. Each item is scored from 1 (not confident at all) to 7 (completely confident). The minimum score is 7 and the maximum score is 49, and higher scores indicate greater self-efficacy.
Custom-designed barrier self-efficacy questionnaire | Immediately post-intervention (in the intervention group only).
  Confidence in one's ability to overcome the barriers associated with adhering to anti-inflammatory diet. This is a 7-item questionnaire that asks participants how confident they are about overcoming the barriers associated with adhering to the anti-inflammatory diet. Each item is scored from 1 (not confident at all) to 7 (completely confident). The minimum score is 7 and the maximum score is 49, and higher scores indicate greater self-efficacy.
Custom-designed barrier self-efficacy questionnaire | One month post-intervention (for the intervention group and the control group)
  Confidence in one's ability to overcome the barriers associated with adhering to anti-inflammatory diet. This is a 7-item questionnaire that asks participants how confident they are about overcoming the barriers associated with adhering to the anti-inflammatory diet. Each item is scored from 1 (not confident at all) to 7 (completely confident). The minimum score is 7 and the maximum score is 49, and higher scores indicate greater self-efficacy.
Adherence to the anti-inflammatory diet | Baseline (for the intervention group and the control group)
  Participants will complete a 7-day food log. Food logs are then analyzed for the number of servings the participant ate that were approved on the anti-inflammatory diet, the number of servings that were not allowed (cheats) and the total servings eaten over the 7 days. Adherence rates are then determined by calculating [(servings allowed/total servings) * 100].
Adherence to the anti-inflammatory diet | One month post-intervention (for the intervention group and the control group)
  Participants will complete a 7-day food log. Food logs are then analyzed for the number of servings the participant ate that were approved on the anti-inflammatory diet, the number of servings that were not allowed (cheats) and the total servings eaten over the 7 days. These values are then combined to calculate each participant's adherence rate with the formula: [(number of servings eaten that were allowed/total servings eaten) x 100]. Adherence rate will be expressed as a percentage. For example, if the participant ate 50 servings of food over 7 days, with 45 of those servings allowed by the anti-inflammatory diet and 5 servings not allowed (cheats), then the adherence rate would be calculated as: Adherence = 45/50 x 100 Adherence = 90%

SECONDARY OUTCOMES:
Neuropathic pain questionnaire (NPQ) | Baseline (for the intervention group and the control group)
  Neuropathic pain as determined by the Neuropathic Pain Questionnaire (NPQ). The questionnaire consists of 32 items pertaining to three unique categories including sensory items, affective items, and sensitivity items. Sensory items are those related to the specific type and severity of pain felt (e.g., degree of burning, stabbing, throbbing), affective items relate to how the pain affects the participant in daily life (e.g., how irritating is your usual pain?) and sensitivity items related to how various stimuli may act to increase pain (e.g., increased pain due to heat). Participants are asked to rate their pain for each item numerically on a scale from 0-100 whereby 0 indicated the complete absence of pain and 100 indicated the worst pain imaginable. Scores from each of the three categories are averaged. Thus, the minimum score for each category is 0 and the maximum score for each category is 100, which higher scores indicating worse pain.
Neuropathic pain questionnaire (NPQ) | One month post-intervention (for the intervention group and the control group)
  Neuropathic pain as determined by the Neuropathic Pain Questionnaire (NPQ). The questionnaire consists of 32 items pertaining to three unique categories including sensory items, affective items, and sensitivity items. Sensory items are those related to the specific type and severity of pain felt (e.g., degree of burning, stabbing, throbbing), affective items relate to how the pain affects the participant in daily life (e.g., how irritating is your usual pain?) and sensitivity items related to how various stimuli may act to increase pain (e.g., increased pain due to heat). Participants are asked to rate their pain for each item numerically on a scale from 0-100 whereby 0 indicated the complete absence of pain and 100 indicated the worst pain imaginable. Scores from each of the three categories are averaged. Thus, the minimum score for each category is 0 and the maximum score for each category is 100, which higher scores indicating worse pain.
Depression as determined by the Centre for Epidemiological Studies depression (CES-D) questionnaire | Baseline (for the intervention group and the control group)
  Depression as determined by the Centre for Epidemiological Studies depression (CES-D) This is a 20-item questionnaire that asks participants to rate their depressive symptoms over the last 7 days, and each item is scored from 0-3. The minimum score for the questionnaire 0 and the maximum score is 60, with higher scores indicating worse depressive symptomology. Any score above 15 is indicative of clinical depression, but should not be taken as a diagnosis by itself.
Depression as determined by the Centre for Epidemiological Studies depression (CES-D) questionnaire | One month post-intervention (for the intervention group and the control group)
  Depression as determined by the Centre for Epidemiological Studies depression (CES-D) This is a 20-item questionnaire that asks participants to rate their depressive symptoms over the last 7 days, and each item is scored from 0-3. The minimum score for the questionnaire 0 and the maximum score is 60, with higher scores indicating worse depressive symptomology. Any score above 15 is indicative of clinical depression, but should not be taken as a diagnosis by itself.

CONTACTS AND LOCATIONS:
Overall Officials: David S Ditor, PhD, Principal Investigator — Brock University
Locations (1):
- Brock University, St. Catharines, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
Available upon reasonable request to the Principal Investigator